CLINICAL TRIAL: NCT03936738
Title: Posttraumatic Stress Disorder and Quality of Life of Avalanche Survivors From 2014 to 2018, Based on the French North Alpine Avalanche Register: Risk Factor Analysis
Brief Title: Posttraumatic Stress Disorder and Quality of Life of Avalanche Survivors From 2014 to 2018, Based on the French North Alpine Avalanche Register
Acronym: ESPTAvalanche
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC19.033; 2018-A02942-53 (Other: ID RCB)
Record Dates: First submitted 2019-04-18; First posted 2019-05-03 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Post Traumatic Stress Disorder; Avalanche, Landslide, or Mudslide; Quality of Life
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to identify if an avalanche accident has a psychological impact on avalanche victims.

The investigators hypothesize that being exposed to an avalanche could generate enough stress to develop posttraumatic stress symptoms or even more, an authentic posttraumatic stress disorder (PTSD). Additionally, the investigators think that such symptoms might lead to physical and psychological distress in daily life. Lastly, the investigators suppose that a serious traumatism, a complete and/or prolonged burial, the death of a family member or a closed friend could be a potential risk factors to develop PTSD symptoms in avalanche victims. To evaluate post traumatic stress symptoms and the quality of life of avalanche survivors, the investigators use the Impact of Event Scale - Revised and the Short Form 12. These two scales are included in a standardized questionnaire, which is submitted to avalanche victims during a phone call.

DETAILED DESCRIPTION:
It is already known that a traumatism, whatever nature or gravity, could lead to acute stress symptoms and a posttraumatic stress disorder (PTSD) one month after (1). In the last decades, less than ten studies showed that avalanche survivors are likely to develop PTSD, even sixteen years after exposure (2, 3). In those studies, authors focused on natural disaster avalanches (on habitations or roads). This study would like to evaluate psychological impact of an avalanche accident occurring during mountain recreational activities.

The primary outcome concerns the research of PTSD symptoms using the Impact of Event Scale - Revised (IES-R). It is a 22 items scale, which explores specifics symptoms of Post Traumatic Stress Disorder that may have occurred during the week before the interview. It concerns 3 different possible areas of PTSD: intrusion (eight items), avoidance (eight items) and hyperarousal symptoms (six items). Each item ranges from 0 (not at all) to 4 (extremely). The total score of the IES-R ranges between 0 and 88. A score equal or more than 33 is highly in favour of PTSD (91% sensitivity, 82% specificity, 90% positive predictive value and 84% negative predictive value). However, above 33 the diagnostic of posttraumatic stress disorder must be confirmed by a psychiatric analysis. Our results will be separated in two categories for the analysis: 1) IES-R score higher or equal to 33; 2) IES-R score lower than 33.

The secondary outcome is the result of the Short Form 12 questionnaire (SF-12). The SF-12 consists of 12 items selected from the "Medical Outcomes Study 36-items Short-Form Health Survey" (SF-36) to reproduce the Physical Component Summary and Mental Component Summary scales in the general US population. The SF-12 Health Survey was developed in the United States to provide a shorter alternative to the SF-36. The SF-12 contains a subset of 12 items from the SF-36, including one or two items from each of the eight SF-36 scales (general health, physical role, physical bodily, vitality, social and emotional functioning, role emotional and mental health). SF-12 Physical and Mental Components are scored from 0 to 100. A higher score indicates a better health state. Scores will be compared to literature data.

Study population concerns avalanche survivors in the French Northern Alps during the last four years. Furthermore, the investigators will try to identify risk factors to develop PTSD in these circumstances. They will try to know if survivors have changed their mountain practice after the accident. From 2014 to 2018, there were 211 avalanche victims in the French North Alps included in the North Alpine Avalanche Register (RENAAV), 132 victims survived. Considering the rate of non-response, the investigators are expecting between 50 to 80 subjects to be analysed. Data will be collected in the medical records and during a phone interview with a standardized questionnaire. A rate of 9,2 % of posttraumatic stress symptoms is expected, corresponding to the prevalence of PTSD (1) after traumatism.

Concerning statistical analysis, quantitative data will be described in terms of mean, standard deviation, median and extreme values. Qualitative data will be described in terms of absolute frequency and percentage by modality. The 95% confidence intervals will be presented. Quantitative data will be compared by a Student's parametric test, replaced by the Wilcoxon test in case of deviation from the normality of distribution. Categorical data will be compared by a Chi 2 test or Fischer's exact test in case of too small sample. A threshold of significance will be retained for a value of p < 0.05. Univariate and multivariate analyses will be performed to independently identify risk factors at a higher frequency of PTSD.

The research team received the approval of ethical research committees since the March 19th of 2019.

ELIGIBILITY:
Inclusion Criteria:

* Adults men and women involved in an avalanche in the French North Alps from the 1rs of December 2014 to 31th of May 2018
* Non opposed during the phone call

Exclusion Criteria:

* Age < 18, when the avalanche occurred
* Non French speaking persons
* Victims deprived of their liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects exposed to an avalanche in the French North Alps and included in the North Alpine Avalanche Register (RENAAV) from the 1st of December 2014 to the 31th of May 2018.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Prospective evaluation of the prevalence of Posttraumatic Stress Disorder of the avalanche survivors included in the RENAAV from December 2014 to May 2018. | Data will be gathered by phone from May to June 2019, all interviews will be conducted in the same place by the same person. Subjects will be randomly contacted.
  The primary outcome is the total score obtained to the Impact of Event Scale Revised (IES-R). This score is validated, translated in french, easy and fast to achieve during a phone call. It is a 22 questions scale which explore the three categories of posttraumatic stress symptoms : intrusion, avoidance, and hyperarousal. Total score ranges between 0 and 88. Results will be separated into three categories : 1) score higher than or equal to 33 ; 2) score between 12 to 32 ; and 3) score lower than or equal to 11. We choose a cut-off score of 33 as seen in the literature. Above 33, the diagnostic of posttraumatic stress disorder must be confirmed with a psychiatric analysis (sensibility = 91 %, specificity = 87 %).

SECONDARY OUTCOMES:
Evaluation of the quality of life, physical and psychological health of an avalanche survivor included in the RENAAV. | Data will be gathered by phone from May to June 2019, all interviews will be conducted in the same place by the same person. Subjects will be randomly contacted.
  The secondary outcome is the result of the Short Form 12 questionnaire (SF-12). The SF-12 consists of 12 items selected from the "Medical Outcomes Study 36-items Short-Form Health Survey" (SF-36) to reproduce the Physical Component Summary and Mental Component Summary scales in the general US population. The SF-12 Health Survey was developed in the United States to provide a shorter alternative to the SF-36. The SF-12 contains a subset of 12 items from the SF-36, including one or two items from each of the eight SF-36 scales (general health, physical role, physical bodily, vitality, social and emotional functioning, role emotional and mental health). SF-12 Physical and Mental Components are scored from 0 to 100. A higher score indicates a better health state. Scores will be compared to literature data.
Analysis of risk factors associated with the onset of Post Traumatic Stress disorder (PTSD) symptoms. | Data will be gathered by phone from May to June 2019, all interviews will be conducted in the same place by the same person. Subjects will be randomly contacted.
  To do this analyse, we form two groups : those who have a Impact of Event Scale Revised (IES-R) score higher than or equal to 33 (PTSD +) ; and those who have a score lower tha 33 (PTSD -).
  The following risk factors will be analysed :
  * Demographic data : age, sex, family and professional situation
  * Severity of physical trauma (calculated with the Injury Severity Scale)
  * Cardiac arrest at extraction time
  * Complete or partial burial
  * Short or prolonged burial
  * Death of a person in the accident
  * Lost of family member or closed friend
  * Length of stay in Intensive care unit
  * Medical history of previous traumatism
  * Psychiatrical history
  * Psychiatric or psychologic care immediately after the accident
  * Medical treatment by anti psychotic, and antidepressant drug after the accident
  * Mountain activity practiced when the accident occurred
  * Outing accompanied by a mountain professional
Research of mountain practice changing. | Data will be gathered by phone from May to June 2019, all interviews will be conducted in the same place by the same person. Subjects will be randomly contacted.
  Three questions will be answered concerning mountain practice, at the end of the interview : Do they currently practice the mountain activity they were doing when avalanche occurred ? How long after the accident ? Did they acquired new mountain security geers (such as airbag backpack, avalanche transceiver, snow probe and shovel). The statistical analysis will be descriptive for this section.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble Alpes, Grenoble, France

REFERENCES:
- [Result] Breslau N. The epidemiology of trauma, PTSD, and other posttrauma disorders. Trauma Violence Abuse. 2009 Jul;10(3):198-210. doi: 10.1177/1524838009334448. Epub 2009 Apr 30. PMID 19406860
- [Result] Thordardottir EB, Valdimarsdottir UA, Hansdottir I, Resnick H, Shipherd JC, Gudmundsdottir B. Posttraumatic stress and other health consequences of catastrophic avalanches: A 16-year follow-up of survivors. J Anxiety Disord. 2015 May;32:103-11. doi: 10.1016/j.janxdis.2015.03.005. Epub 2015 Mar 28. PMID 25935315
- [Result] Parry-Jones B, Parry-Jones WL. Post-traumatic stress disorder: supportive evidence from an eighteenth century natural disaster. Psychol Med. 1994 Feb;24(1):15-27. doi: 10.1017/s0033291700026799. PMID 8208880
- [Result] Johnsen BH, Eid J, Lovstad T, Michelsen LT. Posttraumatic stress symptoms in nonexposed, victims, and spontaneous rescuers after an avalanche. J Trauma Stress. 1997 Jan;10(1):133-40. doi: 10.1023/a:1024820716613. PMID 9018684
- [Result] Finnsdottir T, Elklit A. Posttraumatic sequelae in a community hit by an avalanche. J Trauma Stress. 2002 Dec;15(6):479-85. doi: 10.1023/A:1020969906251. PMID 12482187
- [Derived] Leonard C, Charriau-Perret A, Debaty G, Belle L, Ricard C, Sanchez C, Dupre PM, Panoff G, Bougerol T, Viglino D, Blancher M; Northern French-Alps Emergency Network ("RENAU"). Survivors of avalanche accidents: posttraumatic stress disorder symptoms and quality of life: a multicentre study. Scand J Trauma Resusc Emerg Med. 2021 Jul 19;29(1):96. doi: 10.1186/s13049-021-00912-3. PMID 34281606